CLINICAL TRIAL: NCT06432218
Title: A Randomized Controlled Trial of the Effectiveness of Patient Education in the Clinical Management of Pessary
Brief Title: Patient Education in the Clinical Management of Pessary
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Peking University People's Hospital (Other); Shandong University (Other); Tongji Hospital (Other); Third Military Medical University (Other); Changsha Hospital for Maternal and Child Health Care (Other); Hangzhou Women's Hospital (Unknown); Shenzhen People's Hospital (Other); Foshan Women's and Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: K5558
Record Dates: First submitted 2024-05-10; First posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the conventional education plus video education group (Experimental): Watch video as well as receive conventional guidance.
  Interventions: Other: video education; Other: conventional education
- the conventional education group (Active Comparator): Receive conventional guidance.
  Interventions: Other: conventional education

INTERVENTIONS:
Other: video education — A re-watchable video provided before pessary fitting which mainly includes a short introduction of pessary treatment for pelvic organ prolapse, tips and tricks for wearing and self-management of pessary, possible adverse reactions and remedy.
  Arms: the conventional education plus video education group
Other: conventional education — Conventional verbal/paper instruction and counseling from a specialized doctor or nurse before pessary fitting.

SUMMARY:
This study is a prospective, randomized, controlled, single-blinded, multi-center clinical trial. Symptomatic patients with pelvic organ prolapse (POP) stage II, III or IV arranged to undergo pessary treatment will be randomized into either the experimental group or the control group. All patients will receive conventional verbal/paper instruction and counseling from a specialized doctor or nurse before pessary fitting, and the experimental group will receive additional patient education in the form of a re-watchable video. The video mainly includes a short introduction of pessary treatment for pelvic organ prolapse, tips and tricks for wearing and self-management of pessary, possible adverse reactions and remedy. All patients will receive regular pessary fitting and be followed up for 1 year. Self-assessment questionnaires will be used to assess the patients' willingness to pessary treatment, anxiety status, treatment satisfaction and efficacy, and to assess the patients' self-management, complications and treatment adherence. Then the differences between the two groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic pelvic organ prolapse of stage II~IV
* Ability to participate in clinical trial and follow-up
* The patient and family understand the study, are willing to participate in the 1-year study, and provide written informed consent

Exclusion Criteria:

* Acute phase of infection of the internal and/or external genital tracts
* Genital fistula
* Suspected or untreated lower genital tract tumors
* Abnormally elevated intra-abdominal pressure (e.g., ascites, tumors)
* Life expectancy less than 1 year
* Cognitive or language communication disorders
* Unable to watch video (e.g., blindness)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Continued usage with satisfaction | 12 months after pessary fitting.
  Continued usage of the pessary and have very much or much improvement in the patient impression of improvement (PGI-I) questionnaire at 1 year.

SECONDARY OUTCOMES:
Knowledge of pessary | Baseline and at pessary fitting.
  Self-rated score from 0 to 10 points (higher scores mean a better outcome).
Willingness to treatment | Baseline, at pessary fitting, and 3 and 12 months after successful pessary fitting.
  Self-rated score from 0 to 10 points (higher scores mean a better outcome).
Anxiety about pessary use | Baseline and at pessary fitting.
  7-item generalized anxiety disorder questionnaire (GAD-7) (the range of scores is 0-21, and higher scores mean a worse outcome), and self-rated score of sleep quality from 0 to 10 points (higher scores mean a better outcome).
Ability to self-manage | 3 and 12 months after successful pessary fitting.
  Self-rated score from 0 to 10 points (higher scores mean a better outcome).
Treatment-related symptoms and complications | 3 and 12 months after successful pessary fitting.
  Self report and physical examination.
Improvement in symptoms | 3 and 12 months after successful pessary fitting.
  Pelvic floor impact questionnaire-7 (PFIQ-7) (the range of scores is 0-300, and higher scores mean a worse outcome)
Improvement in quality of life | 3 and 12 months after successful pessary fitting.
  Pelvic floor distress inventory-20 (PFDI-20) (the range of scores is 0-300, and higher scores mean a worse outcome)
Improvement in sexual activity | 3 and 12 months after successful pessary fitting.
  The pelvic organ prolapse/urinary incontinence sexual questionnaire short form (PISQ-12) (the range of scores is 0-48, and higher scores mean a worse outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Lan Zhu, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No